CLINICAL TRIAL: NCT02513979
Title: The Effect of Angiotensin II Receptor Antagonists on Acute and Chronic Postoperative Pain in Patients Treated for Hypertension.
Brief Title: Postoperative Pain and Angiotensin II Receptor Antagonists
Acronym: PP&ARA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Argyro Fassoulaki, Professor Emeritus, University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHSTSA-102
Record Dates: First submitted 2015-07-28; First posted 2015-08-03 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
Keywords: Angiotensin type II receptor (AT2R) antagonists; Acute postoperative pain; Chronic postoperative pain; Abdominal surgery
MeSH Terms: conditions — Hypertension; Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- angiotensin type II receptor antagonists (Active Comparator): Hypertensive patients treated with angiotensin type II receptor antagonists
  Interventions: Drug: Angiotensin type II receptor antagonists
- No treatment (No Intervention): Normotensive patients

INTERVENTIONS:
Drug: Angiotensin type II receptor antagonists — Angiotensin type II receptor antagonists given to hypertensive patients treated with high blood pressure
  Other Names: AT2R antagonists
  Arms: angiotensin type II receptor antagonists

SUMMARY:
An angiotensin II type 2 receptor (AT2R) antagonist has been assessed for its efficacy in neuropathic pain with promising results. A considerable number of patients undergoing surgery under general anesthesia are hypertensive and receive drugs to control high blood pressure, including angiotensin II receptor antagonists. These drugs may attenuate the acute and/or chronic postoperative pain or decrease the analgesic requirements after surgery. The aim of the present study is to assess the early postoperative pain and analgesic requirements in patients treated with antagonists of the angiotensin II receptors for at least three months before surgery compared to normotensive patients.

DETAILED DESCRIPTION:
Patients ASA I-III, aged between 35 and 79 years old, with BMI ≤ 35, scheduled for abdominal surgery, thus gynecological, urological and general surgery procedures will be recruited for the study. All patients will be scheduled in the morning list, informed for the study and will be asked to give written informed consent.

Exclusion Criteria will be patients on analgesic, antidepressive, or sedative consumption during the previous one month, mental impairment, not speaking Greek or refusing to give written informed consent, diabetics, patients receiving antihypertensive treatment other than angiotensin type II receptor (AT2R) antagonists.

Two groups of patients will be stydied: Patients hypertensive (the hypertensive group) receiving treatment for blood pressure control with angiotensin II receptor antagonists for at least three months preoperatively and a normotensive group.

Measurements

* Pain intensity (visual analogue scale: VAS) from 0 to 100 will be reported 2, 4, 8, and 24 hours postoperatively with 0 representing no pain and 100 excruciate worst pain. Pain will be recorded at rest and subsequently patients will be asked to cough for three times.
* Analgesics consumed at the same time points will be recorded.
* Patient satisfaction (VAS 0-100) 24 h postoperatively (with special reference to pain)
* Three months postoperatively patients will be contacted by phone and will be asked if they experience pain related to surgery or not. If yes pain characteristics, thus burning, pricking etc. will be recorded.
* Three months postoperatively patients will be asked whether they used analgesics after discharge from the hospital for the postoperative pain.

Statistics Primary outcome of the study: Pain intensity 24 hours postoperatively after cough in patients receiving angiotensin II receptor antagonists, or no antihypertensive therapy. Secondary outcomes of the study are pain intensity 2, 4, 8 and 24 hours postoperatively at rest, 2, 4 and 8 hours after cough, analgesic consumption , 2, 4, 8 and 24 hours postoperatively, patient satisfaction regarding pain, presence of pain three months after surgery and if present its characteristics. Also, analgesic consumption during the first three months postoperatively due to surgery.

Statistics Power analysis: A 30% difference in pain intensity after cough 24 hours postoperatively between the angiotensin II receptor antagonists treated group compared and the treated group.

Acute pain at rest and after cough all the time points as defined by the study design will be compared between patients receiving antihypertensive treatment (angiotensin II receptors antagonists) and the controls.

Cumulative analgesics consumed 2, 4, 8 and 24 hours after surgery will be compared between the two groups.

The presence of chronic postsurgical pain and the need or not of analgesic intake due to chronic pain three months after surgery will be also compared between the hypertensive treated and normotensive patients.

Parametric or non-parametric tests will be used for normal and no normal distributions respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 35 and 79 years
* ASA II or III
* BMI ≤ 35
* Elective abdominal surgery Exclusion Criteria:-
* Patients on analgesic, antidepressive, or sedative consumption during the last month
* Mental impairment
* Not speaking fluently Greek language
* Refuse to give written informed consent
* Diabetics
* Patients receiving antihypertensive treatment other than angiotensin type II receptor (AT2R) antagonists

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Acute pain after cough | 24 hours postoperatively
  Intensity of pain after cough measured with the Visual Analogue Scale (VAS 0-100 mm)

SECONDARY OUTCOMES:
Acute pain at rest | 2, 4, 8 and 24 hours postoperatively
  Intensity of pain at rest measured with the Visual Analogue Scale (VAS 0-100 mm)
Acute pain after cough | 2, 4 and 8 hours postoperatively
  Intensity of pain after cough measured with the Visual Analogue Scale (VAS 0-100 mm)
Analgesic consumption | 2, 4, 8 and 24 hours postoperatively
  All analgesics converted to morphine equivalent (mg)
Chronic pain | Three months postoperatively
  Present or absent, if present characteristics (pricking, burning, throbbing)
Analgesic consumption for chronic pain | Three months postoperatively
  Yes or not, number of pills

OTHER OUTCOMES:
Patient satisfaction | 24 hours postoperatively
  Patient satisfaction measured in a 0-100 mm scale with special reference to postoperative pain management

CONTACTS AND LOCATIONS:
Overall Officials: Argyro Fassoulaki, MD, Principal Investigator — Aretaieio University Hospital; Marianna Zotou, MD, Study Director — St Savas Hospital
Locations (1):
- Argyro Fassoulaki, Athens, Greece